CLINICAL TRIAL: NCT01784549
Title: A Multi-center Phase II Randomized Study of Customized Neoadjuvant Therapy Versus Standard Chemotherapy in Non-small Cell Lung Cancer (NSLC) Patients With Resectable Stage IIIA (N2) Disease (CONTEST-TRIAL)
Brief Title: Customized Neoadjuvant Versus Standard Chemotherapy in NSCL Patients With Resectable Stage IIIA (N2)Disease
Acronym: CONTEST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Collaborators: Azienda Sanitaria Locale di Cagliari (Other); Azienda Ospedaliera San Gerardo di Monza (Other); Ospedale Santa Croce-Carle Cuneo (Other); Azienda Ospedaliera S. Maria della Misericordia (Other); Istituto Tumori Giovanni Paolo II, BARI (Unknown); Azienda Ospedaliera dei Colli Monaldi-Cotugno-CTO, Napoli (Unknown); Azienda Ospedaliera Santa Maria Degli Angeli (Other); Azienda Ospedaliera San Camillo Forlanini (Other); Azienda Ospedaliera San Giovanni Battista (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); Azienda Sanitaria Locale n.2 Savonese (Other); ASL TO4, Chivasso (Unknown); Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento (Other); Istituto Clinico Humanitas (Other); Azienda Ospedaliera "Sant'Andrea" (Other); Azienda Ospedaliera, Ospedale Civile di Legnano (Other); Azienda Ospedaliera Spedali Riuniti di Livorno, Livorno (Unknown)
Responsible Party: Principal Investigator, Francesco Grossi, Chief, Lung Cancer Unit, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONTEST TRIAL RF-2009-1530324; 2011-005267-24 (EudraCT Number)
Record Dates: First submitted 2013-02-02; First posted 2013-02-06 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCL; biomarkers; Customized Neoadjuvant Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin Docetaxel (Active Comparator): - Cisplatin + Docetaxel day 1 q 21 days for 3 cycles
  Interventions: Drug: Cisplatin Docetaxel Gefitinib Pemetrexed Vinorelbine Gemcitabine
- Gefitinib Pemetrexed Vinorelbine Gemcitabine (Experimental): * Gefitinib day for 8 wks;
  * Pemetrexed day 1 q 21 days for 3 cycles;
  * Docetaxel day 1 + Vinorelbine days 1,8 q 21 days for 3 cycles;
  * Docetaxel days 1,8 + Gemcitabine days 1,8 q 21 days for 3 cycles;
  * Cisplatin + Docetaxel day 1 q 21 days for 3 cycles;
  * Cisplatin day 1+ Gemcitabine days 1,8 q 21 days for 3 cycles;
  Interventions: Drug: Cisplatin Docetaxel Gefitinib Pemetrexed Vinorelbine Gemcitabine

INTERVENTIONS:
Drug: Cisplatin Docetaxel Gefitinib Pemetrexed Vinorelbine Gemcitabine

SUMMARY:
* The investigators hypothesized that NSCL patients receiving therapy based on their baseline tumor markers levels would attain higher response rates than patients in the control arm receiving non customized therapy.
* patients with stage IIIA(N2) NSCLC will be randomized in a 2:1 ratio to customized therapy based on biomarkers status (ERCC1, RRM1, TS and EGFR mutation) vs standard chemotherapy.
* The primary objective of this multicenter trial is to compare pathological complete response of all subjects randomized, by treatment arm.
* Secondary objectives are to compare all randomized subjects by treatment arm for: response rate, disease-free survival, overall survival, one, two and three year survival and safety profile.

The study is expected to demonstrate both the feasibility of this approach and the logistic problems associated with a biomarker-driven therapeutic strategy in NSCLC.

DETAILED DESCRIPTION:
- Subjects will be stratified by histology and biological markers (ERCC1, RRM1, TS, EGFR mutation). Randomization will be centralized at the coordinating centre site. Patients will receive chemotherapy with cisplatin + docetaxel or customized therapy for 3 cycles (60 days with gefitinib) before surgery.

Every 4 months for 3 years and then every 6 months for 2 years following surgery, subjects will be assessed by the investigator for adverse events related to study drug, documentation of post study therapies received, DFS, and survival.

- Periodic evaluations of the trial data will be conducted by an independent data monitoring committee to ensure subject safety and the validity and scientific merit of the study.

Assuming that the study is not stopped at the planned futility analyses or for safety reasons, the final analysis will take place after the targeted number of events (pathological complete response) is reached, which is estimated to take place 24 months post study initiation.

- The pathological complete response (pCR)in the two groups will be computed in the ITT populations and compared by means of the chi-square test without continuity correction. For exploratory purposes, a multivariate logistic regression model will be fitted to the data, with the pCR as the response variable and treatment (standard/ experimental) and histo/molecular subgroup as covariate. The heterogeneity of the relative efficacy of the tailored approach in the various subgroups (=subgroup analysis) will be evaluated by including in the model the appropriate set of treatment-by-subgroup interaction terms, using the standard likelihood ratio test. Time-to-event analyses (DFS and OS) will use standard Kaplan-Meier estimators (with the Log-rank test) and semi-parametric PH regression models. Safety will be summarized based on adverse events, vital signs and laboratory assessments. A group sequential design is used to compare the Overall Survival in the two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a signed and dated written informed consent document prior to any study specific procedures.
* Age ≥18 years, male or female.
* Histologically confirmed NSCLC.
* Specimen tumor tissue obtained from mediastinoscopy
* ECOG Performance status (PS) 0-1.
* Stage IIIA(N2) patients with technical operable disease limited to T1a,b, T2a,b N2 M0; T3 (>7 cm) N2 M0.
* Medically fit for resection by lobectomy or pneumonectomy.
* Radiologically measurable disease (RECIST v1.1 criteria).
* Prior surgery for NSCLC if resected ≥5 years.
* No prior chemotherapy, targeted-therapy, investigational therapy or radiation for NSCLC.
* No uncontrolled medical problems.
* No superior vena cava syndrome.
* Peripheral neuropathy must be ≤ grade 1.
* Acceptable hematologic and chemistry parameters.
* Creatinine clearance >50 ml/min.
* Female patients or their partners must be surgically sterile or be postmenopausal, or agree to use effective contraception while in trial treatment and for 3 months thereafter.
* Female patients with reproductive potential must have a negative pregnancy test (serum or urine) within 72 hours prior to starting treatment.
* Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures including patient reported measures.

Exclusion Criteria:

* Any evidence of mixed histology including elements of small cell or carcinoid lung cancer.
* Stage IIIA patients limited to T3 N1 M0; T3 (invasion) N2 M0; T4 N0, N1 M0.
* Any clinically significant GI abnormalities, which may impair intake, transit or absorption of gefitinib, such as the inability to take oral medication.
* Current enrollment in another therapeutic clinical trial.
* Any psychiatric or cognitive disorder that would limit the understanding or rendering of informed consent and/or compromise compliance with the requirements of this study.
* Past medical history of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease
* Pre-existing idiopathic pulmonary fibrosis evidence by computerized tomography (CT) scan at baseline.
* Uncontrolled or significant CV disease, including: myocardial infarction within 12 months; uncontrolled angina within 6 months; congestive heart failure within 6 months; diagnosed or suspected congenital long QT syndrome;
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes);
* Prolonged QTc interval on pre entry ECG.
* Any history of second or third degree heart block (may be eligible if currently have a pacemaker);
* Heart rate <50/minute on baseline ECG;
* Uncontrolled hypertension.
* Evidence of prior malignancy (other than non melanoma skin cancer or in situ cervical cancer, or localized and presumed cured prostate cancer with PSA < ULN) within the last 3 years.
* Other severe acute or chronic medical condition that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator.
* Patients in whom corticosteroid premedication was contraindicated.
* HIV-positive patients on active treatment.
* Medications are prohibited at baseline and prior to randomization if they affect the pharmacokinetics of gefitinib, cisplatin, docetaxel, gemcitabine, vinorelbine and pemetrexed or if they are mainly metabolized by CYP3A4.
* Patients who are otherwise eligible can be enrolled only if drug substitution is performed with acceptable clinical outcome prior to enrollment: known severe hypersensitivity to gefitinib or other chemotherapeutic agents or any of the excipients of the products.
* Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response | 30 days

SECONDARY OUTCOMES:
Overall Survival (OS) | at 1, 2, and 5 years
Disease-Free Survival (DFS) | at 1, 2, and 5 years
Overall Response (OR) | at 1, 2, and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Grossi, MD, Principal Investigator — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (1):
- IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy